CLINICAL TRIAL: NCT02936414
Title: Berberine Effect on Cytokine, CRP, Metabolic Disturbance as an Adjunctive Therapy in Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ber-2015-TJAH
Record Dates: First submitted 2016-09-29; First posted 2016-10-18 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-10

CONDITIONS: Schizophrenia
Keywords: Berberine; Cytokine; CRP; Metabolism; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Berberine; Coptidis rhizoma extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Berberine group (Experimental): Berberine (300 mg/tid), as an adjuvant therapy will be used on the basis of the SGAs monotherapy.
  Interventions: Drug: Berberine
- Placebo group (Placebo Comparator): Accept placebo(300 mg/tid)+SGAs monotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — Berberine (300 mg/tid), as an adjuvant therapy will be used on the basis of the SGAs monotherapy.
  Other Names: Huang Liansu; Rhizoma coptidis
  Arms: Berberine group
Drug: Placebo — Accept placebo(300 mg/tid)+SGAs monotherapy.
  Arms: Placebo group

SUMMARY:
The etiology and pathogenesis of schizophrenia remains unclear. Immune dysfunction hypothesis for schizophrenia has attracted increasing attention of the researchers, substantial evidences suggested the levels of C-reaction protein and cytokine such as IL-1β, IL-6, TNF-α markedly elevated in patients with schizophrenia which may be particularly relevant for the cognitive impairment and metabolic disturbance of schizophrenia. In recent years, it has been demonstrated the beneficial effects of berberine on regulating lipid and glucose metabolism, reducing the proinflammatory status and improving cognition. As the investigators known, the report of berberine being used in schizophrenia is rare. This protocol is aim to evaluate berberine, as an adjunctive therapy, on inflammatory markers, lipid and glucose metabolism, cognition in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who age 18 to 60 years diagnose schizophrenia according the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID).
* The patients have illness for less than 5 years and have stable dose of the current antipsychotic drug for at least one month.
* Well established compliance with inpatient treatment per treating clinician's judgment. On baseline, at least 60 for Positive and Negative Syndrome Scale (PANSS) total score.
* Able to complete the cognitive assessment battery Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods during the study.

Exclusion Criteria:

* Individuals who refuse to provide informed consent.
* Currently substance abuse or psychiatrically unstable per treating clinician's judgment.
* One with significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases also not suitable for this trial.
* Currently on anti-inflammatory or immunosuppressant medication including oral steroids and history of chronic infection (including tuberculosis, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition pregnancy or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The change of glucose | Change from Baseline Glucose at 12 weeks
The change of insulin | Change from Baseline insulin at 12 weeks
The change of HbA1c | Change from Baseline HbA1c at 12 weeks
The change of lipid profile | Change from Baseline lipid profile at 12 weeks
The change of CRP | Change from Baseline CRP at 12 weeks
The change of IL-1β | Change from Baseline IL-1β at 12 weeks
The change of IL-6 | Change from Baseline IL-6 at 12 weeks
The change of TNF-α | Change from Baseline TNF-α at 12 weeks
The change of Cognitive function assessed with The MATRICS Consensus Cognitive Battery (MCCB) | Change from Baseline Cognitive function at 12 weeks
  The MATRICS Consensus Cognitive Battery (MCCB) for Cognitive function

SECONDARY OUTCOMES:
The change of clinical symptoms assessed with The Positive and Negative Syndrome Scale | Change from Baseline clinical symptoms at 12 weeks
  The Positive and Negative Syndrome Scale for clinical symptoms
Adverse event | At 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No